CLINICAL TRIAL: NCT03495661
Title: Uppsala Spinal Stenosis Study
Brief Title: Decompression vs Physical Training for the Treatment of Lumbar Spinal Stenosis
Acronym: UppSten
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: u1
Record Dates: First submitted 2018-03-22; First posted 2018-04-12 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Spinal Stenosis; Spinal Stenosis Lumbar; Degeneration Lumbar Spine; Degeneration Spine; Neurogenic Claudication Co-Occurrent and Due to Spinal Stenosis of Lumbar Region; Pseudoclaudication Syndrome
Keywords: lumbar spine stenosis; decompression; laminectomy; physiotherapy; physical therapy; electroneurography; ENG; electromyography; EMG; Neurogenic Claudication; Pseudoclaudication
MeSH Terms: conditions — Spinal Stenosis | interventions — Decompression; Laminectomy

STUDY DESIGN:
Intervention Model Description: prospective clinical randomised clinical trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical (Decompression) (Active Comparator): Central decompression of the stenotic segment(s) with undercutting of the lateral recesses.
  Interventions: Procedure: Decompression
- Non-surgical (No Intervention): Physical therapy according to the "Östersund model": training on stationary bicycle 30 min, 3 times/week under 4 months.

INTERVENTIONS:
Procedure: Decompression — Central decompression of the stenotic segment(s) with undercutting of the lateral recesses.
  Other Names: Laminectomy
  Arms: Surgical (Decompression)

SUMMARY:
Lumbar spinal stenosis (LSS) is characterized by low back and leg pain, walking disturbances and sometimes instability, impaired balance and numbness of the lower limbs. This condition is caused by degenerative changes in the lumbar spine including bulging discs, osteophytes from the arthritic facet joints and thickened ligamentum flavum which together cause narrowing of the spinal canal and thus affect the lumbar nerve roots. This diagnosis is attracting more and more interest due to the aging population with increasing demands for physical activity. LSS is the most common indication for spinal surgery. The surgical treatment involves relieving the pressure from the nerve structures in the stenotic segments through a posterior approach. In several studies, surgery has been shown to have better results than the conservative treatment. However, methodological difficulties and a large proportion of cross-over in these studies indicate that there is still uncertainty about whether surgery is generally a better option.

It has been speculated whether the compression of the nerve roots causes in some patients permanent nerve damage with muscle denervation, while in other cases a reinnervation and recovery of the function may occur. Results from neurography and EMG studies have been shown these modalities to have a possible predictive value for the natural process of LSS. If a neurophysiological examination could be able to predict which patients are able to benefit from surgery, many patients could avoid surgery and the risks involved in it.

The aim of this study is primarily to evaluate whether surgery with decompression leads to superior results than the non-surgical treatment with structured physical therapy.

The main secondary aim is to investigate by means of Neurography and EMG, whether the degree of neurological affection caused by nerve compression affects the outcome of surgery for LSS.

DETAILED DESCRIPTION:
Background

Lumbar spinal stenosis (LSS) is characterized by low back and leg pain, walking disturbances and sometimes instability, impaired balance and numbness of the lower limbs. This condition is caused by degenerative changes in the lumbar spine including bulging discs, osteophytes from the arthritic facet joints and thickened ligamentum flavum which together cause narrowing of the spinal canal and thus affect the lumbar nerve roots. LSS affects mainly older populations and is unusual under 50 years old. This diagnosis is attracting more and more interest due to the aging population with increasing demands for physical activity. LSS is the most common indication for spinal surgery. The surgical treatment involves relieving the pressure from the nerve structures in the stenotic segments through a posterior approach. The hypertrophic ligaments and parts of the facet joints are removed (i.e., decompression). Adding fusion to the decompression for stabilization of the decompressed segment has not been shown to provide superior results than decompression alone. In several studies, surgery has been shown to have better results than the conservative treatment. However, methodological difficulties and a large proportion of cross-over in these studies indicate that there is still uncertainty about whether surgery is generally a better option.

After decompression, only 60-70% of patients reported to be satisfied with the result and a minor proportion of them experienced even no improvement at all [Strömqvist]. Conservative treatment has shown in some studies to have good results for some patient groups and other studies have shown that the benefit of the surgical treatment decreases over time and that physical exercise may reduce the need for surgery. Moreover, surgery itself has a positive placebo effect that can improve symptoms in some diseases.

It has been speculated whether the compression of the nerve roots causes in some patients permanent nerve damage with muscle denervation, while in other cases a reinnervation and recovery of the function may occur. Results from neurography and EMG studies have been shown these modalities to have a possible predictive value for the natural process of LSS. If a neurophysiological examination could be able to predict which patients are able to benefit from surgery, many patients could avoid surgery and the risks involved in it.

The degeneration of the lumbar spine is progressively impairing the spinal sagittal balance. The need to make extensive correction and fusion in addition to the decompression in order to restore the sagittal balance is debated among spinal surgeons. The experience gained from previous RCTs is that the patients' back pain is reduced by decompression only. Many patients also report that their posture improved after decompression alone.

Previous trials in the connective tissue and blood samples have shown that proinflammatory factors and nociceptors (molecules that induce pain) are upregulated in patients with patellar tendinosis which is an inflammatory condition. Changes in the connective tissue that cause LSS are mainly inflammatory (arthritic facet joints and ligamentum flavum) and a possible theory around LSS pathophysiology may be that the nerves are biologically affected by proinflammatory factors and nociceptors. Identification of some of these factors could lead to better explanation of the pathomechanism behind the nerve compression in LSS and to the development of future pharmacological treatments to be used in conjunction with surgery.

Aims

The aim of this study is primarily to evaluate whether surgery with decompression leads to superior results than the non-surgical treatment with structured physical therapy. For this evaluation, the Oswestry Disability Index (ODI) will be used.

The main secondary aim is to investigate by means of Neurography and EMG, whether the degree of neurological affection caused by nerve compression affects the outcome of surgery for LSS.

Aims The aim of this study is primarily to evaluate whether surgery with decompression leads to superior results than the non-surgical treatment with structured physical therapy. For his evaluation, the Oswestry Disability Index (ODI) will be used.

The main secondary aim is to investigate by means of Neurography and EMG, whether the degree of neurological affection caused by nerve compression affects the outcome of surgery for LSS.

The questions at issue are:

1. Does decompression provide a better clinical outcome than the non-surgical treatment?
2. Is there any correlation between the clinical grade of symptoms and the degree of neurological affection measured by ENG/EMG?
3. Is there any connection between the neurological affection and the proinflammatory markers/nociceptors in the blood as well as in histological findings from ligamentum flavum? Are these correlated with the clinical grade of symptoms?
4. Does decompression provide superior neurological recovery, measured by ENG/EMG, in comparison to the non-surgical treatment ?
5. Can decompression improve the spinal sagittal balance?

Follow-up 6 months, 1, 2 and 5 years

The results at 2 years will be the most important goal of the study, on which the main clinical results will be built. The neurophysiological results can be analyzed and presented after the 6-month follow up.

Flow-chart

Recruitment The patient is recruited during an outpatient visit to a surgeon. Oral and written information about the study is given.

ICF The patient gives oral and written consent. The consent is documented in the patient journal and the written consent is filed in the study document binder.

Baseline data - PROMs via Swespine Study

* 6MWT
* Scoliosis standing digital X-rays (AP and lateral views)
* ENG/EMG
* Blood samples for analysis of inflammatory markers (OLINK)

Randomizing Simple block randomization to the two treatment arms.

Treatment arms A. Decompression. Central decompression of the stenotic segments with undercutting of the lateral recesses, free mobilization, and routine follow-up postoperatively by physiotherapist.

B. Non-surgical treatment. Exercise on exercise bike according to the "Östersund model" [Nord] 30 min, 3 times/week for 4 months.

Follow-up 6 months - PROMs via Swespine Study

* 6MWT
* Scoliosis standing digital X-rays (AP and lateral views)
* ENG/EMG
* Blood samples for analysis of inflammatory markers (OLINK)

Cross-over Feasibility for cross-over from group B till A after 6-month follow-up.

Follow-up 1,2 years - PROMs via Swespine Study

- 6MWT

Follow -up 5 years - PROMs via Swespine Study

In the treatment group A, in conjunction with the surgical procedure, ligamentum flavum will be collected (which is usually removed during the decompression surgery) and will be examined with histological methods regarding proinflammatory markers and nociceptors . An 1x1 cm tissue piece will be dissected and saved. The ligament samples will be examined by immunohistochemistry and with proteomics analysis. Proteomics analysis will be performed in collaboration with Olink Uppsala (www.olink.com) where 92 inflammation-related factors will be investigated. Sample management will be in accordance with the Ethics Examination Act of Human Research (2003: 460) and according to the rules of Uppsala Biobank.

ELIGIBILITY:
Inclusion criteria

1. Age 50-85 years.
2. Clinical symptoms of lumbar spinal stenosis (pseudoclaudication) that indicate and motivate surgery. NRS in lower limbs ≥3.
3. MRI with finding of LSS at 1-3 lumbar levels. Dural sac area ≤ 75 mm² or degree of stenosis C or D according to Schizas classification.
4. The surgical treatment to be provided is decompression alone.
5. The patient has given oral and written informed consent to the participation in the study.

Exclusion criteria

1. Degenerative deformity with Cobb angle > 20°.
2. Spondylolysis.
3. Symptomatic osteoarthritis in the lower limbs that affects and limits their function.
4. Arterial insufficiency (claudication intermittent) .
5. Past lumbar surgery other than disc hernia.
6. Conditions that affect the spine such as ankylosing spondylitis, Diffuse Idiopathic Skeletal Hyperostosis (DISH), spondylodiscitis/infections, malignancy, neurological diseases.
7. Heart and lung diseases that present a significant risk for surgery or make it impossible for the patient to take part in physical training program (ASA>3).
8. Polyneuropathies.
9. Psychological factors that make the patient incapable of inclusion in the study (eg drug addiction, dementia)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline
  Through the Swedish National Spine Registry (SweSpine)
Oswestry Disability Index (ODI) | 6 months
  Through the Swedish National Spine Registry (SweSpine)
Oswestry Disability Index (ODI) | 1 year
  Through the Swedish National Spine Registry (SweSpine)
Oswestry Disability Index (ODI) | 2 years
  Through the Swedish National Spine Registry (SweSpine)
Oswestry Disability Index (ODI) | 5 years
  Through the Swedish National Spine Registry (SweSpine)

SECONDARY OUTCOMES:
Motor Amplitude (ENG) | Baseline and 6 months postoperatively
Denervation Activity (EMG) | Baseline and 6 months follow-up
Sensory Amplitude (ENG) | Baseline and 6 months follow-up
Late Responses (F-wave and H.Reflex) | Baseline and 6 months follow-up
Motor Unit Number Index (MUNIX) | Baseline and 6 months follow-up
Grade of Reinnervation (EMG) | Baseline and 6 months follow-up
EQ-5D | Baseline and 6 months, 1, 2, 5 years follow-up
  Through the Swedish National Spine Registry (SweSpine)
NRS for Low Back and Leg Pain | Baseline and 6 months, 1, 2, 5 years follow-up
  Through the Swedish National Spine Registry (SweSpine)
Subjective Walking Ability | Baseline and 6 months, 1, 2, 5 years follow-up
  Through the Swedish National Spine Registry (SweSpine)
Global Assessment (GA) | Baseline and 6 months, 1, 2, 5 years follow-up
  Through the Swedish National Spine Registry (SweSpine)
Patient Satisfaction | Baseline and 6 months, 1, 2, 5 years follow-up
  Through the Swedish National Spine Registry (SweSpine)
Objective Walking Ability | Baseline and 6 months, 1, 2 years follow-up
  6 Minutes Walk Test (6MWT)
Lumbar Lordosis (LL) and Sagittal Vertebral Axis (SVA) | Baseline and 6 months follow-up
  Standing Scoliosis X-rays (AP and Lateral view)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Pazarlis, MD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Pazarlis K, Punga A, Schizas N, Sanden B, Michaelsson K, Forsth P. Study protocol for a randomised controlled trial with clinical, neurophysiological, laboratory and radiological outcome for surgical versus non-surgical treatment for lumbar spinal stenosis: the Uppsala Spinal Stenosis Trial (UppSten). BMJ Open. 2019 Aug 20;9(8):e030578. doi: 10.1136/bmjopen-2019-030578. PMID 31434781

DOCUMENTS (1):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT03495661/Prot_000.pdf